CLINICAL TRIAL: NCT05765240
Title: Comparison of the Effects of Topical Hyaluronic Acid and Laser Application on Healing in Children After Tooth Extraction
Brief Title: The Effects of Topical Hyaluronic Acid and Laser Application on Wound Healing in Children
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Atlas University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2015-KAEK-43-19-25
Record Dates: First submitted 2023-03-01; First posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-02

CONDITIONS: Wound Heal; Tooth Extraction Status Nos

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (Experimental): Hyaluronic acid gel will be applied to the extraction site of the patients in group 1 immediately after the extraction.
  Interventions: Drug: Hyaluronic Acid Topical Gels
- Group 2 (Experimental): Alveolar socket in group 2, will ve irradiated with an energy dose of J/cm2, 20mW/670 nm potency and 4 for 7 minutes immediately after extraction.
  It will be irradiated with an energy dose of J/cm2.
  Interventions: Procedure: Diode Laser Biostimulation
- Control Group (No Intervention)

INTERVENTIONS:
Drug: Hyaluronic Acid Topical Gels — Hyaluronic acid is a linear polysaccharide found naturally in different organs and tissues such as the extracellular matrix of connective tissue, synovial fluid, embryonic mesenchyme, and skin. The periodontal ligament is a key element found in periodontal tissues such as the gingiva, alveolar bone, and cementum. It plays a regulatory role in the inflammatory response, impedes the penetration of viruses and bacteria into the tissue, and is involved in inflammation, granulation tissue formation, epithelial formation, and tissue remodeling. There are no reported drug interactions or contraindications for the use of hyaluronic acid.
  Arms: Group 1
Procedure: Diode Laser Biostimulation — Laser therapy can amplify wound healing by increasing cell regeneration and modulating the immune response. In animal experiments with diode laser, it was observed that postoperative low-level laser application increased wound healing. Diode laser applied at frequencies of 20 mW and 670 nm and 200 mW and 820 nm accelerated clot organization and new vessel formation after tooth extraction.
  Arms: Group 2

SUMMARY:
Tooth extraction is one of the major surgical procedures that can cause dental anxiety and dental fear in pediatric patients as a result of traumatic experiences. Preventing pain and infection by appropriate means during and after this application increases patient comfort and helps to develop patient cooperation for possible future dental experiences.

In the current literature, it has been shown that topical hyaluronic acid applications have a role in reducing infection and pain.

There are also studies in the literature showing that tissue biostimulation with different doses of diode laser application accelerates wound healing by promoting cell regeneration.

Although there are studies showing that two different applications accelerate wound healing, there is no study comparing the effectiveness of these two methods. In addition, there is no study evaluating extraction wound healing in pediatric patients.

Our study will be the first to evaluate tooth extraction wound healing in pediatric patients and to compare these two methods.

DETAILED DESCRIPTION:
Sample Size:

Our study will include 60 children aged between 5-13 years who are systemically healthy and volunteer to participate in the study, with indications for extraction of primary or permanent molars for various reasons.

In the study, the GPOWER 3.1 package program was used to determine the sufficient sample volume.

Steps followed when calculating sample volume;

1st type margin of error (α) = 0.05 The mean (1.72) and standard deviation (1.14) values of the 7th day VAS scores of the participants in the "control" group were taken into account.

The mean (0.92) and standard deviation (0.81) values of the 7th day VAS scores of the participants in the "Hyaluronic Acid (HA)" group were taken into account.

Using the relevant mean and standard deviation values, the effect size was calculated as 0.9876543.

The power of the test was taken as (1-β) = 0.80. As a result of the calculations, the sample volume that will provide the power of the test (1-β) = 0.80 was determined as 54 people in total, with a minimum of 18 in each group.

Considering the possible reductions in the follow-up process, the sample number was determined as 60 people, 20 people in each group.

Study Design:

Children with primary or permanent molar extraction indications will be divided into three as:

Group 1: Hyaluronic Acid Gel Group Group 2: Diode Laser Group The control group.

As a result of clinical and radiographic examination, the extraction of primary or permanent molar teeth will be performed by a single investigator under local anesthesia.

All patient groups will be evaluated by a single investigator at the time of the extraction and on the 7th, 14th, and 21st days following the extraction. The same investigator will perform an intraoral examination before extraction and record the caries status using DMFT and dft scoring.

Pain assessment will be made through the Wong-Baker Faces Pain Scale suitable for ages 3-18. The patient will be asked to score the pain felt at the extraction site during the period between follow-up appointments, and a total of 3 assessments will be made.

In all groups, the presence of edema and infection will be evaluated by a single investigator on the 7th, 14th, and 21st days following the extraction.

Wound dimensions (dehiscent, mesiodistal and buccolingual longest distances on the socket) will be determined by a single investigator immediately after the extraction and on the 3rd, 7th, and 14th days following the extraction, and recorded with photographs taken from a standard distance.

In the control group, the wound area will be followed without any application after tooth extraction.

Hyaluronic acid gel will be applied to the extraction site of the patients in the hyaluronic acid gel group immediately after the extraction.

In the diode laser group, the alveolar socket will be irradiated with a potency of 20mW/670 nm and an energy dose of 4 J/cm2 for 7 minutes immediately after extraction.

ELIGIBILITY:
Inclusion Criteria:

Being systemically healthy

Having at least one primary or permanent molar extraction indication

The fact that at least 1/3 of the primary tooth root with an extraction indication has not been resorbed

Have not used antibiotics in the last 6 months

Exclusion Criteria:

Presence of systemic disease

Deciduous teeth with highly resorbed roots

Use of antibiotics in the last 6 months

-

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-27 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Wound healing | One month
  Healing index of Landry will be used

SECONDARY OUTCOMES:
Post-operative pain | Two weeks
  VAS pain scale data and number of painkillers used (if any) will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Atlas University, Istanbul, Kağıthane, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided